CLINICAL TRIAL: NCT00458341
Title: A Phase 2 Study of PTC124 as an Oral Treatment for Nonsense-Mutation-Mediated Cystic Fibrosis
Brief Title: A Study of Ataluren in Pediatric Participants With Cystic Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PTC Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PTC124-GD-006-CF
Record Dates: First submitted 2007-04-06; First posted 2007-04-10 (Estimated); Results first posted 2020-03-06 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-02

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis; Nonsense mutation; Premature stop codon
MeSH Terms: conditions — Cystic Fibrosis | interventions — ataluren

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ataluren 4, 4, and 8 mg/kg, then ataluren 10, 10, and 20 mg/kg (Experimental): During Cycle 1, participants will receive ataluren at 4 mg/kg in the morning, 4 mg/kg at midday, and 8 mg/kg in the evening for 14 days, followed by a 14-day follow-up period without treatment. Then, the participants will crossover to the other ataluren dose regimen (ataluren 10, 10, and 20 mg/kg) for Cycle 2.
  Interventions: Drug: Ataluren
- Ataluren 10, 10, and 20 mg/kg, then ataluren 4, 4, and 8 mg/kg (Experimental): During Cycle 1, participants will receive ataluren at 10 mg/kg in the morning, 10 mg/kg at midday, and 20 mg/kg in the evening for 14 days, followed by a 14-day follow-up period without treatment. Then, the participants will crossover to the other ataluren dose regimen (ataluren 4, 4, and 8 mg/kg) for Cycle 2.
  Interventions: Drug: Ataluren

INTERVENTIONS:
Drug: Ataluren — Ataluren will be provided as a vanilla-flavored powder to be mixed with water, milk, or apple juice. Participants are to receive a total of 42 doses of ataluren during each cycle, for a total of 84 doses of ataluren in both cycles.
  Other Names: PTC124

SUMMARY:
In some participants with cystic fibrosis (CF), the disease is caused by a nonsense mutation (premature stop codon) in the gene that makes the cystic fibrosis transmembrane regulator (CFTR) protein. Ataluren has been shown to partially restore CFTR production in animals with CF due to a nonsense mutation. The main purpose of this study is to understand whether ataluren can safely increase functional CFTR protein in the cells of participants with CF due to a nonsense mutation.

DETAILED DESCRIPTION:
In this study, participants with CF due to a nonsense mutation will be treated with a new investigational drug called ataluren. Evaluation procedures (history, physical examination, blood and urine tests to assess organ function, electrocardiogram [ECG], chest x-ray, and CF-specific tests) to determine if a participant qualifies for the study will be performed within 21 days prior to the start of treatment. Eligible participants with nonsense-mutation-mediated CF will receive 2 repeated 28-day cycles, each comprising of 14 days on therapy and 14 days off therapy. In a crossover design, participants will be randomized to receive ataluren treatment in Cycle 1 by either of the following regimens:

* Ataluren, given 3 times per day (TID) with a regimen of 4 milligrams/kilograms (mg/kg) at breakfast, 4 mg/kg at lunch, and 8 mg/kg at dinner, or
* Ataluren, given 3 TID with a regimen of 10 mg/kg at breakfast, 10 mg/kg at lunch and 20 mg/kg at dinner.

In Cycle 2, participants will then receive the drug according to the regimen opposite from that given in Cycle 1.

There will be a 2-night stay at the clinical research center at the beginning and at the end of each 14 days of ataluren treatment, which means that there will be four 2-night stays at the clinical research center during the study. During the study, ataluren efficacy, safety, and pharmacokinetics (PK) will be evaluated periodically with measurements of transepithelial potential difference (TEPD), nasal mucosal brushing to assess for cellular CFTR messenger ribonucleic acid (mRNA) and protein, medical history, physical examinations, blood tests, sputum test, urinalysis, ECGs, chest x-ray, and pulmonary function tests.

The measurement of TEPD, also known as nasal potential difference, provides a sensitive evaluation of sodium and chloride transport directly in secretory epithelial cells. TEPD assessments are made on the nasal epithelium cells lining the inferior turbinate because these cells are easier to access than the respiratory epithelial cells lining the lower airways and have been shown to have the same ion transport characteristics. As an endpoint, TEPD has the advantage that it can detect chloride transport changes that are a quantitative integration of the presence, functional activity, and apical location of the CFTR in airway cells. Furthermore, it is a direct measure of CFTR activity that is not likely to be affected by supportive or palliative treatments for CF (with the possible exception of systemically administered aminoglycoside antibiotics).

ELIGIBILITY:
Inclusion Criteria: Participants must meet all of the following conditions to be eligible for enrollment into the study:

1. Diagnosis of CF based on conclusively abnormal sweat test (sweat chloride >35 milliequivalents [mEq]/liter).
2. Abnormal nasal epithelial TEPD total chloride conductance (a more electrically negative value than 5 mV for Δchloride-free+isoproterenol).
3. Presence of a mutation in both alleles.
4. Documentation that a blood sample has been drawn for reconfirmation of the presence of a nonsense mutation in the CFTR gene.
5. Age ≥6 years.
6. Body weight ≥25 kg.
7. FEV1 ≥40% of predicted for age, gender, and height.
8. Oxygen saturation ≥92% on room air.
9. Willingness of male and female participants, if not surgically sterile, to abstain from sexual intercourse or employ a barrier or medical method of contraception during the study drug administration and follow-up periods.
10. Negative pregnancy test (for females of childbearing potential).
11. Willingness and ability to comply with scheduled visits, drug administration plan, study procedures (including TEPD measurements, clinical laboratory tests, pulmonary function tests, and PK sampling), and study restrictions.
12. Ability to provide written informed consent and/or assent.
13. Evidence of signed and dated informed consent document (by the participant or a legal guardian) indicating that the participant and/or the legal guardian has been informed of all pertinent aspects of the trial.

Exclusion Criteria: The presence of any of the following conditions will exclude a participant from enrollment in the study:

1. Prior exposure to ataluren.
2. Prior or ongoing medical condition (for example, concomitant illness, alcoholism, drug abuse, psychiatric condition), medical history, physical findings, ECG findings, or laboratory abnormality that, in the Investigator's opinion, could adversely affect the safety of the participant, makes it unlikely that the course of treatment or follow-up would be completed, or could impair the assessment of study results.
3. Ongoing acute illness including acute upper or lower respiratory infections within 2 weeks before start of study treatment.
4. History of major complications of lung disease (including recent massive hemoptysis or pneumothorax) within 2 months prior to start of study treatment.
5. Abnormalities on screening chest x-ray suggesting clinically significant active pulmonary disease other than CF, or new, significant abnormalities such as atelectasis or pleural effusion which may be indicative of clinically significant active pulmonary involvement secondary to CF.
6. Positive hepatitis B surface antigen, hepatitis C antibody test, or human immunodeficiency virus (HIV) test.
7. Hemoglobin <10 grams/deciliter (g/dL).
8. Serum albumin <2.5 g/dL.
9. Abnormal liver function (serum total bilirubin > the upper limit of normal, or serum alanine aminotransferase (ALT), aspartate aminotransferase (AST), or gamma-glutamyl transferase (GGT) >2.0 times the upper limit of normal).
10. Abnormal renal function (serum creatinine >1.5 times upper limit of normal).
11. Pregnancy or breast-feeding.
12. History of solid organ or hematological transplantation.
13. Exposure to another investigational drug within 14 days prior to start of study treatment.
14. Ongoing participation in any other therapeutic clinical trial.
15. Ongoing use of thiazolidinedione peroxisome proliferator-activated receptor gamma (PPAR γ) agonists, for example, rosiglitazone (Avandia® or equivalent) or pioglitazone (Actos® or equivalent).
16. Change in intranasal medications (including use of corticosteroids, cromolyn, ipratropium bromide, phenylephrine, or oxymetazoline) within 14 days prior to start of study treatment.
17. Change in treatment with systemic or inhaled corticosteroids within 14 days prior to start of study treatment.
18. Use of or requirement for inhaled gentamicin or amikacin within 14 days prior to start of study treatment or during study treatment.
19. Requirement for systemic aminoglycoside antibiotics within 14 days prior to start of study treatment.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2007-03-23 (Actual); Primary Completion 2008-02-29 (Actual); Study Completion 2008-02-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Sermet-Gaudelus, MD, Principal Investigator — Hopital Necker
Locations (3):
- Belgium (2):
  - Reine Fabiola Hospital, Brussels
  - UZ Gasthuisberg Leuven, Leuven
- Hopital Necker Enfants Malades, Paris, France

REFERENCES:
- [Derived] Sermet-Gaudelus I, Boeck KD, Casimir GJ, Vermeulen F, Leal T, Mogenet A, Roussel D, Fritsch J, Hanssens L, Hirawat S, Miller NL, Constantine S, Reha A, Ajayi T, Elfring GL, Miller LL. Ataluren (PTC124) induces cystic fibrosis transmembrane conductance regulator protein expression and activity in children with nonsense mutation cystic fibrosis. Am J Respir Crit Care Med. 2010 Nov 15;182(10):1262-72. doi: 10.1164/rccm.201001-0137OC. Epub 2010 Jul 9. PMID 20622033

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized so that half received the lower-dose level in Cycle 1 and then the higher-dose level in Cycle 2 (low-to-high dose sequence) and half received the higher-dose level in Cycle 1 and then the lower-dose level in Cycle 2 (high-to-low dose sequence).
Groups:
- Ataluren 4, 4, and 8 mg/kg, Then Ataluren 10, 10, and 20 mg/kg: During Cycle 1, participants received ataluren at 4 milligrams (mg/kg) in the morning, 4 mg/kg at midday, and 8 mg/kg in the evening for 14 days, followed by a 14-day follow-up period without treatment. Then, the participants crossed over to the other ataluren dose regimen (ataluren 10, 10, and 20 mg/kg) for Cycle 2.
- Ataluren 10, 10, and 20 mg/kg, Then Ataluren 4, 4, and 8 mg/kg: During Cycle 1, participants received ataluren at 10 mg/kg in the morning, 10 mg/kg at midday, and 20 mg/kg in the evening for 14 days, followed by a 14-day follow-up period without treatment. Then, the participants crossed over to the other ataluren dose regimen (ataluren 4, 4, and 8 mg/kg) for Cycle 2.
Period: Cycle 1
Arm/Group | Ataluren 4, 4, and 8 mg/kg, Then Ataluren 10, 10, and 20 mg/kg | Ataluren 10, 10, and 20 mg/kg, Then Ataluren 4, 4, and 8 mg/kg
Started (Cycle 1: from first dose of PTC124 through day before first dosing date in Cycle 2.) | 15 | 15
Received at Least 1 Dose of Study Drug | 15 | 15
Completed | 14 (1 participant did not complete Cycle 1 since all procedures were not performed due to adverse event.) | 15
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Cycle 2
Arm/Group | Ataluren 4, 4, and 8 mg/kg, Then Ataluren 10, 10, and 20 mg/kg | Ataluren 10, 10, and 20 mg/kg, Then Ataluren 4, 4, and 8 mg/kg
Started (Cycle 2: first dosing date after 2-week rest period in Cycle 1 through end-of-study follow-up.) | 15 (The participant who did not complete Cycle 1 was eligible for Cycle 2 and completed Cycle 2.) | 15
Received at Least 1 Dose of Study Drug | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of study drug.
Groups:
- Ataluren 4, 4, and 8 mg/kg, Then Ataluren 10, 10, and 20 mg/kg: During Cycle 1, participants received ataluren at 4 mg/kg in the morning, 4 mg/kg at midday, and 8 mg/kg in the evening for 14 days, followed by a 14-day follow-up period without treatment. Then, the participants crossed over to the other ataluren dose regimen (ataluren 10, 10, and 20 mg/kg) for Cycle 2.
- Total: Total of all reporting groups
Arm/Group | Ataluren 4, 4, and 8 mg/kg, Then Ataluren 10, 10, and 20 mg/kg | Ataluren 10, 10, and 20 mg/kg, Then Ataluren 4, 4, and 8 mg/kg | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 12 (3.53) | 13 (3.38) | 12.5 (3.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 9 | 7 | 16

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Chloride Transport at Day 14 of Cycles 1 and 2
Description: Nasal transepithelial potential difference (TEPD) was assessed in each participant using standardized techniques. Warmed solutions of Ringer's solution, amiloride, chloride-free gluconate, isoproterenol, and adenosine triphosphate (ATP) were perfused for ≥3-minute sequentially through a nasal catheter while a voltage tracing was recorded. Total chloride transport was computed for each nostril. The total chloride transport values were calculated by subtracting the voltages at the end of a perfusion from the voltage at the end of an earlier perfusion (isoproterenol - amiloride). The average of the values for each nostril was computed. If the assessment was available in only 1 nostril, this value was used as if it were the average of both nostrils. Baseline data for Cycle 1 and Cycle 2 and change from Baseline data at Day 14 of Cycles 1 and 2 are presented.
Time Frame: Baseline of Cycle 1 and Cycle 2, Day 14 of Cycle 1 and Cycle 2 (1 cycle=28 days)
Population: All randomized participants who received at least 1 dose of study drug and had evaluable chloride transport data.
Measure: Mean (Standard Deviation); unit: millivolts (mV)
Arm/Group | Ataluren 4, 4, and 8 mg/kg, Then Ataluren 10, 10, and 20 mg/kg | Ataluren 10, 10, and 20 mg/kg, Then Ataluren 4, 4, and 8 mg/kg
Number analyzed (Participants) | 15 | 15
millivolts (mV)
  Baseline of Cycle 1 | 1.45 (5.671) | 0.66 (4.563)
  Change at Day 14 of Cycle 1: number analyzed (Participants) | 14 | 14
  Change at Day 14 of Cycle 1 | -2.81 (6.543) | -2.69 (7.289)
  Baseline of Cycle 2: number analyzed (Participants) | 15 | 13
  Baseline of Cycle 2 | -0.92 (4.474) | -3.76 (6.729)
  Change at Day 14 of Cycle 2: number analyzed (Participants) | 14 | 13
  Change at Day 14 of Cycle 2 | -2.39 (5.426) | 1.10 (7.179)
Statistical Analysis 1: Comparison: Ataluren 4, 4, and 8 mg/kg, Then Ataluren 10, 10, and 20 mg/kg; Baseline of Cycle 1 versus Day 14 of Cycle 1; Test type: Other; p = 0.133, t-test, 2 sided — Threshold for significance at 0.05 level
Statistical Analysis 2: Comparison: Ataluren 10, 10, and 20 mg/kg, Then Ataluren 4, 4, and 8 mg/kg; Baseline of Cycle 1 versus Day 14 of Cycle 1; Test type: Other; p = 0.190, t-test, 2 sided — Threshold for significance at 0.05 level
Statistical Analysis 3: Comparison: Ataluren 4, 4, and 8 mg/kg, Then Ataluren 10, 10, and 20 mg/kg; Baseline of Cycle 2 versus Day 14 of Cycle 2; Test type: Other; p = 0.123, t-test, 2 sided — Threshold for significance at 0.05 level
Statistical Analysis 4: Comparison: Ataluren 10, 10, and 20 mg/kg, Then Ataluren 4, 4, and 8 mg/kg; Baseline of Cycle 2 versus Day 14 of Cycle 2; Test type: Other; p = 0.592, t-test, 2 sided — Threshold for significance at 0.05 level

2. Primary Outcome: Number of Participants With a Chloride Transport Response at Day 14 of Cycles 1 and 2
Description: Nasal TEPD was assessed in each participant using standardized techniques. Warmed solutions of Ringer's solution, amiloride, chloride-free gluconate, isoproterenol, and ATP were perfused for ≥3-minute sequentially through a nasal catheter while a voltage tracing was recorded. Total chloride transport was computed for each nostril. The total chloride transport values were calculated by subtracting the voltages at the end of a perfusion from the voltage at the end of an earlier perfusion (isoproterenol - amiloride). The average of the values for each nostril was computed. If the assessment was available in only 1 nostril, this value was used as if it were the average of both nostrils. Response to study treatment defined as an increase in total chloride transport as indicated by a change of at least -5 mV in nasal TEPD.
Time Frame: Day 14 of Cycle 1 and Cycle 2 (1 cycle=28 days)
Population: All randomized participants who received at least 1 dose of study drug and had evaluable chloride transport response data.
Measure: Count of Participants; unit: Participants
Arm/Group | Ataluren 4, 4, and 8 mg/kg, Then Ataluren 10, 10, and 20 mg/kg | Ataluren 10, 10, and 20 mg/kg, Then Ataluren 4, 4, and 8 mg/kg
Number analyzed (Participants) | 15 | 15
Participants
  Day 14 of Cycle 1: number analyzed (Participants) | 14 | 14
  Day 14 of Cycle 1 | 4 | 4
  Day 14 of Cycle 2: number analyzed (Participants) | 14 | 13
  Day 14 of Cycle 2 | 4 | 2
Statistical Analysis 1: Comparison: Ataluren 4, 4, and 8 mg/kg, Then Ataluren 10, 10, and 20 mg/kg; Analysis of Cycle 1 data. Analysis was to compare the observed rate with the null hypothesis response rate of 10%; Test type: Other; p = 0.021, Chi-squared
Statistical Analysis 2: Comparison: Ataluren 10, 10, and 20 mg/kg, Then Ataluren 4, 4, and 8 mg/kg; Analysis of Cycle 1 data. Analysis was to compare the observed rate with the null hypothesis response rate of 10%; Test type: Other; p = 0.021, Chi-squared
Statistical Analysis 3: Comparison: Ataluren 4, 4, and 8 mg/kg, Then Ataluren 10, 10, and 20 mg/kg; Analysis of Cycle 2 data. Analysis was to compare the observed rate with the null hypothesis response rate of 10%; Test type: Other; p = 0.021, Chi-squared
Statistical Analysis 4: Comparison: Ataluren 10, 10, and 20 mg/kg, Then Ataluren 4, 4, and 8 mg/kg; Analysis of Cycle 2 data. Analysis was to compare the observed rate with the null hypothesis response rate of 10%; Test type: Other; p = 0.518, Chi-squared

3. Primary Outcome: Number of Participants With Normalization of Chloride Transport Between Baseline and Day 14 of Cycles 1 and 2
Description: Nasal TEPD was assessed in each participant using standardized techniques. Warmed solutions of Ringer's solution, amiloride, chloride-free gluconate, isoproterenol, and ATP were perfused for ≥3-minute sequentially through a nasal catheter while a voltage tracing was recorded. Total chloride transport was computed for each nostril. The total chloride transport values were calculated by subtracting the voltages at the end of a perfusion from the voltage at the end of an earlier perfusion (isoproterenol - amiloride). The average of the values for each nostril was computed. If the assessment was available in only 1 nostril, this value was used as if it were the average of both nostrils. Normalization of chloride transport (normal range [NR]) was defined as nasal TEPD that was at least as electrically negative as -5 mV. Normalization in chloride transport can also be referred to as hyperpolarization.
Time Frame: Overall Baseline and Day 14 of Cycle 1 and Cycle 2 (1 cycle=28 days)
Population: All randomized participants who received at least 1 dose of study drug and had evaluable normalization of chloride transport data.
Measure: Count of Participants; unit: Participants
Arm/Group | Ataluren 4, 4, and 8 mg/kg, Then Ataluren 10, 10, and 20 mg/kg | Ataluren 10, 10, and 20 mg/kg, Then Ataluren 4, 4, and 8 mg/kg
Number analyzed (Participants) | 14 | 14
Participants
  Within NR at Baseline of Cycle 1 | 0 | 0
  Within NR at Day 14 of Cycle 1 | 1 | 5
  Outside NR at Baseline/in NR at Day 14 of Cycle 1 | 1 | 5
  Within NR at Baseline of Cycle 2: number analyzed (Participants) | 14 | 13
  Within NR at Baseline of Cycle 2 | 2 | 4
  Within NR at Day 14 of Cycle 2: number analyzed (Participants) | 14 | 13
  Within NR at Day 14 of Cycle 2 | 6 | 3
  Outside NR at Baseline/in NR at Day 14 of Cycle 2: number analyzed (Participants) | 14 | 13
  Outside NR at Baseline/in NR at Day 14 of Cycle 2 | 6 | 2

4. Secondary Outcome: Change From Baseline in Parameters of Transepithelial Difference at Day 14 of Cycles 1 and 2
Description: To assess TEPD, warmed solutions of Ringer's solution, amiloride, chloride-free gluconate, isoproterenol and ATP were perfused for ≥3-minutes sequentially through a nasal catheter while a voltage tracing was recorded. Total chloride transport was computed per nostril. Totals were calculated by subtracting voltages at end of perfusion from voltage at end of earlier perfusion for: sodium transport (amiloride-Ringer's solution), intrinsic chloride transport (chloride-free gluconate-amiloride), stimulated chloride transport (isoproterenol-chloride-free gluconate), total potential difference (isoproterenol-Ringer's solution), and ATP-mediated chloride transport (ATP-isoproterenol). Basal potential difference voltage was obtained at end of Ringer's solution perfusion. Average values per nostril were computed. If assessment was available in only 1 nostril, the value was used as if it's the average of both nostrils. Baseline data for Cycles 1 and 2 and change from Baseline data are presented.
Time Frame: Baseline of Cycle 1 and Cycle 2, Day 14 of Cycle 1 and Cycle 2 (1 cycle=28 days)
Population: All randomized participants who received at least 1 dose of study drug and had evaluable transepithelial difference data.
Measure: Mean (Standard Deviation); unit: mV
Arm/Group | Ataluren 4, 4, and 8 mg/kg, Then Ataluren 10, 10, and 20 mg/kg | Ataluren 10, 10, and 20 mg/kg, Then Ataluren 4, 4, and 8 mg/kg
Number analyzed (Participants) | 15 | 15
mV
  Basal nasal TEPD, Baseline of Cycle (C)1 | -53.91 (18.81) | -56.51 (20.68)
  Basal nasal TEPD, Change at Day (D)14 of C1: number analyzed (Participants) | 14 | 14
  Basal nasal TEPD, Change at Day (D)14 of C1 | 9.31 (17.72) | -3.70 (13.33)
  Basal nasal TEPD, Baseline of C2: number analyzed (Participants) | 15 | 13
  Basal nasal TEPD, Baseline of C2 | -46.28 (14.46) | -50.02 (17.09)
  Basal nasal TEPD, Change at D14 of C2: number analyzed (Participants) | 14 | 13
  Basal nasal TEPD, Change at D14 of C2 | -6.31 (19.33) | -5.22 (24.48)
  Sodium transport, Baseline of C1 | 34.38 (17.72) | 36.40 (18.44)
  Sodium transport, Change at D14 of C1: number analyzed (Participants) | 14 | 14
  Sodium transport, Change at D14 of C1 | -4.97 (15.30) | 1.55 (18.39)
  Sodium transport, Baseline of C2: number analyzed (Participants) | 15 | 13
  Sodium transport, Baseline of C2 | 28.85 (14.31) | 32.15 (17.72)
  Sodium transport, Change at D14 of C2: number analyzed (Participants) | 14 | 13
  Sodium transport, Change at D14 of C2 | 6.38 (19.81) | 5.50 (20.69)
  Intrinsic chloride transport, Baseline of C1 | 2.38 (4.19) | 1.11 (4.01)
  Intrinsic chloride transport, Change at D14 of C1: number analyzed (Participants) | 14 | 14
  Intrinsic chloride transport, Change at D14 of C1 | -2.54 (4.70) | -2.69 (4.96)
  Intrinsic chloride transport, Baseline of C2: number analyzed (Participants) | 15 | 13
  Intrinsic chloride transport, Baseline of C2 | -1.32 (5.61) | -0.90 (3.44)
  Intrinsic chloride transport, Change at D14 of C2: number analyzed (Participants) | 14 | 13
  Intrinsic chloride transport, Change at D14 of C2 | -1.20 (6.23) | -1.12 (5.34)
  Stimulated chloride transport, Baseline of C1 | -0.93 (2.22) | -0.45 (1.63)
  Stimulated chloride transport, Change at D14 of C1: number analyzed (Participants) | 14 | 14
  Stimulated chloride transport, Change at D14 of C1 | -0.27 (3.44) | 0 (4.26)
  Stimulated chloride transport, Baseline of C2: number analyzed (Participants) | 15 | 13
  Stimulated chloride transport, Baseline of C2 | 0.40 (4.83) | -2.86 (6.98)
  Stimulated chloride transport, Change at D14 of C2: number analyzed (Participants) | 14 | 13
  Stimulated chloride transport, Change at D14 of C2 | -1.19 (5.89) | 2.21 (8.77)
  Total potential difference, Baseline of C1: number analyzed (Participants) | 14 | 15
  Total potential difference, Baseline of C1 | 35.83 (17.25) | 37.06 (17.25)
  Total potential difference, Change at D14 of C1: number analyzed (Participants) | 15 | 14
  Total potential difference, Change at D14 of C1 | -7.77 (12.16) | -1.14 (13.89)
  Total potential difference, Baseline of C2 | 27.93 (15.37) | 28.39 (17.18)
  Total potential difference, Change at D14 of C2: number analyzed (Participants) | 14 | 13
  Total potential difference, Change at D14 of C2 | 3.99 (19.48) | 6.59 (20.20)
  ATP-mediated chloride transport, Baseline C1: number analyzed (Participants) | 11 | 11
  ATP-mediated chloride transport, Baseline C1 | -19.84 (10.22) | -17.65 (10.62)
  ATP-mediated chloride transport, Change at D14, C1: number analyzed (Participants) | 10 | 10
  ATP-mediated chloride transport, Change at D14, C1 | 4.93 (11.56) | -2.95 (15.59)
  ATP-mediated chloride transport, Baseline C2: number analyzed (Participants) | 11 | 10
  ATP-mediated chloride transport, Baseline C2 | -16.87 (13.24) | -16.34 (12.35)
  ATP-mediated chloride transport, Change at D14, C2: number analyzed (Participants) | 9 | 10
  ATP-mediated chloride transport, Change at D14, C2 | -0.38 (17.47) | -4.58 (27.93)

5. Secondary Outcome: Change From Baseline in CFTR Protein in Nasal Mucosa as Determined by Immunofluorescence at Overall Day 56
Description: The immunofluorescence staining of normal epithelial cells (for example, from nasal mucosal curettage) reveals the presence of cystic fibrosis transmembrane regulator (CFTR) protein at the apical surface. Cells were stained with antibodies that recognized an epitope in the C-terminal portion of the CFTR protein, and the cells were imaged microscopically. The percentage of epithelial cells that showed apical CFTR staining was determined by 2 expert readers who were blinded to the timepoint at which the samples were obtained. The scores of the reviewers were averaged to determine the final percentage of cells with apical CFTR. Overall Baseline data for the study and change from overall Baseline data at overall Day 56 are presented.
Time Frame: Overall Baseline, Overall Day 56
Population: All randomized participants who received at least 1 dose of study drug and had evaluable apical cell data.
Measure: Mean (Standard Deviation); unit: percentage of apical cells
Arm/Group | Ataluren 4, 4, and 8 mg/kg, Then Ataluren 10, 10, and 20 mg/kg | Ataluren 10, 10, and 20 mg/kg, Then Ataluren 4, 4, and 8 mg/kg
Number analyzed (Participants) | 15 | 15
percentage of apical cells
  Overall Baseline: number analyzed (Participants) | 12 | 11
  Overall Baseline | 15.95 (16.797) | 10.47 (9.270)
  Change at Overall Day 56: number analyzed (Participants) | 10 | 11
  Change at Overall Day 56 | 10.45 (24.337) | 22.89 (29.389)

6. Secondary Outcome: Change From Baseline in Nonsense Mutation CFTR mRNA in Nasal Mucosa as Determined by Quantitative Real-Time Polymerase Chain Reaction (RT-PCR) Assay at Overall Day 42
Description: The collection and processing of the nasal mucosal curettage from each nostril of each participant for measurement of CFTR protein by immunofluorescence and for quantification of CFTR messenger ribonucleic acid (mRNA) was performed using standardized techniques. The slides were processed and immunostained for detection of CFTR protein. Microscopic images were to be captured photographically for analysis. Because the nasal brushing used to collect nasal mucosal epithelial cells did not result in collection of sufficient cells for RT-PCR to be performed, an insufficient number of paired baseline and follow-up samples were available for analysis. As a result, no data were available to evaluate the effects of ataluren on CFTR mRNA.
Time Frame: Overall Baseline, Overall Day 42
Population: All randomized participants who received at least 1 dose of study drug and had evaluable CFTR mRNA data.
Arm/Group | Ataluren 4, 4, and 8 mg/kg, Then Ataluren 10, 10, and 20 mg/kg | Ataluren 10, 10, and 20 mg/kg, Then Ataluren 4, 4, and 8 mg/kg
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change From Baseline in Pulmonary Function as Measured by Spirometry at Day 14 or 15 of Cycles 1 and 2 and Overall Day 56
Description: Pulmonary function tests, including forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC), and forced expiratory flow25-75 (FEF25-75), were measured using standard spirometry techniques. Overall Baseline data for the study and change from overall Baseline data at Day 14 or 15 of Cycles 1 and 2 and at overall Day 56 are presented.
Time Frame: Overall Baseline, Day 14 or 15 of Cycle 1 and Cycle 2 (1 cycle=28 days), and Overall Day 56
Population: All randomized participants who received at least 1 dose of study drug and had evaluable pulmonary function data.
Measure: Mean (Standard Deviation); unit: percent of predicted
Arm/Group | Ataluren 4, 4, and 8 mg/kg, Then Ataluren 10, 10, and 20 mg/kg | Ataluren 10, 10, and 20 mg/kg, Then Ataluren 4, 4, and 8 mg/kg
Number analyzed (Participants) | 15 | 15
percent of predicted
  FEV1, Overall Baseline | 92.68 (22.645) | 85.14 (27.850)
  FEV1, Change at Day 14 or 15 of Cycle 1: number analyzed (Participants) | 14 | 15
  FEV1, Change at Day 14 or 15 of Cycle 1 | 2.73 (5.848) | -4.60 (7.579)
  FEV1, Change at Day 14 or 15 of Cycle 2 | -0.46 (11.031) | 0.02 (8.801)
  FEV1, Change at Overall Day 56 | -0.36 (12.936) | -0.39 (8.191)
  FVC, Overall Baseline | 101.83 (13.294) | 95.34 (22.515)
  FVC, Change at Day 14 or 15 of Cycle 1: number analyzed (Participants) | 14 | 15
  FVC, Change at Day 14 or 15 of Cycle 1 | 2.52 (7.216) | -2.33 (6.643)
  FVC, Change at Day 14 or 15 of Cycle 2 | -0.44 (7.433) | -0.44 (7.433)
  FVC, Change at Overall Day 56 | -0.65 (9.117) | 1.02 (6.796)
  FEF 25-75%, Overall Baseline | 88.32 (49.740) | 71.20 (41.194)
  FEF 25-75%, Change at Day 14 or 15 of Cycle 1: number analyzed (Participants) | 14 | 15
  FEF 25-75%, Change at Day 14 or 15 of Cycle 1 | 2.98 (19.679) | -3.63 (12.300)
  FEF 25-75%, Change at Day 14 or 15 of Cycle 2 | 3.19 (22.712) | -0.39 (19.192)
  FEF 25-75%, Change at Overall Day 56 | -2.76 (27.406) | -4.29 (23.379)

8. Secondary Outcome: Change From Baseline in Sputum Markers of Inflammation (Free Elastase) at Day 14 or 15 of Cycles 1 and 2 and Overall Day 56
Description: The inflammatory marker free elastase was measured in induced sputum from each participant. Hypertonic saline (3%) inhalation was used to induce the sputum (with efforts made to avoid oropharyngeal contamination). The sputum sample was divided into 4 aliquots (1 aliquot each for determination of cell count, IL-8 level, and elastase activity and 1 aliquot for potential future viscosity measurements). Change from overall Baseline data at Day 14 or 15 of Cycles 1 and 2 and at overall Day 56 are presented.
Time Frame: Overall Baseline, Day 14 or 15 of Cycle 1 and Cycle 2 (1 cycle=28 days), and Overall Day 56
Population: All randomized participants who received at least 1 dose of study drug and had evaluable sputum markers of inflammation data.
Measure: Mean (Standard Deviation); unit: micrograms/milliliters (μg/mL)
Arm/Group | Ataluren 4, 4, and 8 mg/kg, Then Ataluren 10, 10, and 20 mg/kg | Ataluren 10, 10, and 20 mg/kg, Then Ataluren 4, 4, and 8 mg/kg
Number analyzed (Participants) | 15 | 15
micrograms/milliliters (μg/mL)
  Free Elastase, Baseline: number analyzed (Participants) | 12 | 10
  Free Elastase, Baseline | 108.85 (107.617) | 60.92 (56.170)
  Free Elastase, Change at Day 14 or 15 of Cycle 1: number analyzed (Participants) | 10 | 10
  Free Elastase, Change at Day 14 or 15 of Cycle 1 | -37.78 (95.154) | 74.66 (83.258)
  Free Elastase, Change at Day 14 or 15 of Cycle 2: number analyzed (Participants) | 9 | 10
  Free Elastase, Change at Day 14 or 15 of Cycle 2 | -24.40 (93.804) | 37.33 (65.240)
  Free Elastase, Change at Overall Day 56: number analyzed (Participants) | 9 | 10
  Free Elastase, Change at Overall Day 56 | 12.47 (84.427) | 57.18 (139.211)

9. Secondary Outcome: Change From Baseline in Sputum Markers of Inflammation (Matrix Metalloproteinase 9 [MMP-9] Active) at Day 14 or 15 of Cycles 1 and 2 and Overall Day 56
Description: The inflammatory marker MMP-9 active was measured in induced sputum from each participant. Hypertonic saline (3%) inhalation was used to induce the sputum (with efforts made to avoid oropharyngeal contamination). The sputum sample was divided into 4 aliquots (1 aliquot each for determination of cell count, IL-8 level, and elastase activity and 1 aliquot for potential future viscosity measurements). Change from overall Baseline data at Day 14 or 15 of Cycles 1 and 2 and at overall Day 56 are presented.
Time Frame: Overall Baseline, Day 14 or 15 of Cycle 1 and Cycle 2 (1 cycle=28 days), and Overall Day 56
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: nanograms/milliliter (ng/mL)
Arm/Group | Ataluren 4, 4, and 8 mg/kg, Then Ataluren 10, 10, and 20 mg/kg | Ataluren 10, 10, and 20 mg/kg, Then Ataluren 4, 4, and 8 mg/kg
Number analyzed (Participants) | 15 | 15
nanograms/milliliter (ng/mL)
  MMP-9 Active, Baseline: number analyzed (Participants) | 13 | 15
  MMP-9 Active, Baseline | 69431.28 (109894.966) | 20908.56 (28441.612)
  MMP-9 Active, Change at Day 14 or 15 of Cycle 1: number analyzed (Participants) | 11 | 10
  MMP-9 Active, Change at Day 14 or 15 of Cycle 1 | -44527.45 (92493.455) | 71639.89 (150716.037)
  MMP-9 Active, Change at Day 14 or 15 of Cycle 2: number analyzed (Participants) | 11 | 10
  MMP-9 Active, Change at Day 14 or 15 of Cycle 2 | -51330.37 (108057.265) | 14947.54 (69337.080)
  MMP-9 Active, Change at Overall Day 56: number analyzed (Participants) | 10 | 10
  MMP-9 Active, Change at Overall Day 56 | -49644.49 (86334.812) | 56884.39 (158498.793)

10. Secondary Outcome: Change From Baseline in Sputum Markers of Inflammation (Tumor Necrosis Factor-Alpha [TNF-α], Interleukin-8 [IL-8], Transforming Growth Factor Beta 1 [TGF-β1]) at Day 14 or 15 of Cycles 1 and 2 and Overall Day 56
Description: The inflammatory markers TNF-α, IL-8, and TGF-β1 were measured in induced sputum from each participant. Hypertonic saline (3%) inhalation was used to induce the sputum (with efforts made to avoid oropharyngeal contamination). The sputum sample was divided into 4 aliquots (1 aliquot each for determination of cell count, IL-8 level, and elastase activity and 1 aliquot for potential future viscosity measurements). Change from overall Baseline data at Day 14 or 15 of Cycles 1 and 2 and at overall Day 56 are presented.
Time Frame: Overall Baseline, Day 14 or 15 of Cycle 1 and Cycle 2 (1 cycle=28 days), and Overall Day 56
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: picograms/milliliter (pg/mL)
Arm/Group | Ataluren 4, 4, and 8 mg/kg, Then Ataluren 10, 10, and 20 mg/kg | Ataluren 10, 10, and 20 mg/kg, Then Ataluren 4, 4, and 8 mg/kg
Number analyzed (Participants) | 15 | 15
picograms/milliliter (pg/mL)
  IL-8, Baseline: number analyzed (Participants) | 13 | 10
  IL-8, Baseline | 352539.57 (331865.227) | 121879.75 (83684.594)
  IL-8, Change at Day 14 or 15 of Cycle 1: number analyzed (Participants) | 11 | 10
  IL-8, Change at Day 14 or 15 of Cycle 1 | -171764.67 (296343.195) | 98483.55 (154432.714)
  IL-8, Change at Day 14 or 15 of Cycle 2: number analyzed (Participants) | 11 | 10
  IL-8, Change at Day 14 or 15 of Cycle 2 | -71206.95 (289379.557) | -4087.25 (127038.632)
  IL-8, Change at Overall Day 56: number analyzed (Participants) | 10 | 10
  IL-8, Change at Overall Day 56 | -121626.94 (263731.747) | 52880.35 (176223.116)
  TGF-b1, Baseline: number analyzed (Participants) | 12 | 10
  TGF-b1, Baseline | 80.84 (280.044) | 322.56 (612.153)
  TGF-b1, Change at Day 14 or 15 of Cycle 1: number analyzed (Participants) | 9 | 10
  TGF-b1, Change at Day 14 or 15 of Cycle 1 | 0 (0) | -322.56 (612.15)
  TGF-b1, Change at Day 14 or 15 of Cycle 2: number analyzed (Participants) | 10 | 9
  TGF-b1, Change at Day 14 or 15 of Cycle 2 | -97.01 (306.773) | -168.91 (774.276)
  TGF-b1, Change at Overall Day 56: number analyzed (Participants) | 9 | 7
  TGF-b1, Change at Overall Day 56 | -61.32 (367.788) | -392.21 (771.006)
  TNF-alpha, Baseline: number analyzed (Participants) | 11 | 8
  TNF-alpha, Baseline | 203.15 (185.530) | 95.69 (139.550)
  TNF-alpha, Change at Day 14 or 15 of Cycle 1: number analyzed (Participants) | 9 | 8
  TNF-alpha, Change at Day 14 or 15 of Cycle 1 | -58.94 (183.812) | 46.38 (67.679)
  TNF-alpha, Change at Day 14 or 15 of Cycle 2: number analyzed (Participants) | 9 | 8
  TNF-alpha, Change at Day 14 or 15 of Cycle 2 | -85.28 (123.341) | -58.45 (144.728)
  TNF-alpha, Change at Overall Day 56: number analyzed (Participants) | 8 | 8
  TNF-alpha, Change at Overall Day 56 | 1.50 (267.702) | 0.25 (122.285)

11. Secondary Outcome: Change From Baseline in Sputum Markers of Inflammation (Uridine-5'-Triphosphate [UTP]) at Day 14 or 15 of Cycles 1 and 2 and Overall Day 56
Description: The inflammatory marker UTP was measured in induced sputum from each participant. Hypertonic saline (3%) inhalation was used to induce the sputum (with efforts made to avoid oropharyngeal contamination). The sputum sample was divided into 4 aliquots (1 aliquot each for determination of cell count, IL-8 level, and elastase activity and 1 aliquot for potential future viscosity measurements). Change from overall Baseline data at Day 14 or 15 of Cycles 1 and 2 and at overall Day 56 are presented.
Time Frame: Overall Baseline, Day 14 or 15 of Cycle 1 and Cycle 2 (1 cycle=28 days), and Overall Day 56
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: milligrams/deciliter (mg/dL)
Arm/Group | Ataluren 4, 4, and 8 mg/kg, Then Ataluren 10, 10, and 20 mg/kg | Ataluren 10, 10, and 20 mg/kg, Then Ataluren 4, 4, and 8 mg/kg
Number analyzed (Participants) | 15 | 15
milligrams/deciliter (mg/dL)
  UTP, Baseline: number analyzed (Participants) | 13 | 10
  UTP, Baseline | 800.27 (509.794) | 483.31 (222.102)
  UTP, Change at Day 14 or 15 of Cycle 1: number analyzed (Participants) | 11 | 10
  UTP, Change at Day 14 or 15 of Cycle 1 | -202.85 (427.324) | 411.50 (359.669)
  UTP, Change at Day 14 or 15 of Cycle 2: number analyzed (Participants) | 11 | 10
  UTP, Change at Day 14 or 15 of Cycle 2 | -200.94 (549.730) | 198.03 (436.888)
  UTP, Change at Overall Day 56: number analyzed (Participants) | 10 | 9
  UTP, Change at Overall Day 56 | -220.16 (414.258) | -15.86 (242.686)

12. Secondary Outcome: Change From Baseline in Clinically Significant Neutrophil Levels in Blood at Day 14 or 15 of Cycles 1 and 2 and Overall Day 56
Description: To assess inflammatory markers in the blood, neutrophil levels in the blood were measured. Higher levels of neutrophils are indicative of more inflammation. Change from overall Baseline data at Day 14 or 15 of Cycles 1 and 2 and at overall Day 56 are presented.
Time Frame: Overall Baseline, Day 14 or 15 of Cycle 1 and Cycle 2 (1 cycle=28 days), and Overall Day 56
Population: All randomized participants who received at least 1 dose of study drug and had evaluable data of neutrophil levels in blood.
Measure: Mean (Standard Deviation); unit: 10^9/liters
Arm/Group | Ataluren 4, 4, and 8 mg/kg, Then Ataluren 10, 10, and 20 mg/kg | Ataluren 10, 10, and 20 mg/kg, Then Ataluren 4, 4, and 8 mg/kg
Number analyzed (Participants) | 15 | 15
10^9/liters
  Neutrophils - Absolute, Baseline | 3.555 (1.2328) | 4.709 (3.0884)
  Neutrophils - Absolute, Day 14 or 15 of Cycle 1: number analyzed (Participants) | 14 | 15
  Neutrophils - Absolute, Day 14 or 15 of Cycle 1 | -0.332 (1.3416) | -0.330 (2.7710)
  Neutrophils - Absolute, Day 14 or 15 of Cycle 2 | -0.290 (1.4881) | -0.748 (2.2473)
  Neutrophils - Absolute, Overall Day 56 | -0.114 (1.4724) | -0.931 (2.7452)

13. Secondary Outcome: Change From Baseline in Clinically Significant Serum Levels of C-Reactive Protein at Day 14 or 15 of Cycles 1 and 2 and Overall Day 56
Description: To assess inflammatory markers in the blood, serum levels of C-reactive protein were measured. Higher levels of C-reactive protein are indicative of more inflammation. Change from overall Baseline data at Day 14 or 15 of Cycles 1 and 2 and at overall Day 56 are presented.
Time Frame: Overall Baseline, Day 14 or 15 of Cycle 1 and Cycle 2 (1 cycle=28 days), and Overall Day 56
Population: All randomized participants who received at least 1 dose of study drug and had evaluable serum levels of C-reactive data.
Measure: Mean (Standard Deviation); unit: milligrams/liter (mg/L)
Arm/Group | Ataluren 4, 4, and 8 mg/kg, Then Ataluren 10, 10, and 20 mg/kg | Ataluren 10, 10, and 20 mg/kg, Then Ataluren 4, 4, and 8 mg/kg
Number analyzed (Participants) | 15 | 15
milligrams/liter (mg/L)
  C-Reactive Protein, Baseline | 6.432 (4.9133) | 8.273 (7.8838)
  C-Reactive Protein, Day 14 or 15 of Cycle 1: number analyzed (Participants) | 14 | 15
  C-Reactive Protein, Day 14 or 15 of Cycle 1 | -0.150 (1.6337) | 7.059 (16.9563)
  C-Reactive Protein, Day 14 or 15 of Cycle 2 | -0.233 (0.7761) | 2.933 (12.0167)
  C-Reactive Protein, Overall Day 56 | 2.361 (7.4765) | 1.240 (7.7170)

14. Secondary Outcome: Change From Baseline in Body Weight at Day 14 or 15 of Cycles 1 and 2 and Overall Day 56
Description: Body weight were measured for each participant in kilograms (kg). Overall Baseline data for the study and change from overall Baseline data at Day 14 of Cycles 1 and 2 and at overall Day 56 are presented.
Time Frame: Overall Baseline, Day 14 of Cycle 1 and Cycle 2 (1 cycle=28 days), and Overall Day 56
Population: All randomized participants who received at least 1 dose of study drug and had evaluable body weight data.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Ataluren 4, 4, and 8 mg/kg, Then Ataluren 10, 10, and 20 mg/kg | Ataluren 10, 10, and 20 mg/kg, Then Ataluren 4, 4, and 8 mg/kg
Number analyzed (Participants) | 15 | 15
kg
  Overall Baseline | 40.35 (12.239) | 41.72 (11.435)
  Change at Day 14 of Cycle 1: number analyzed (Participants) | 14 | 15
  Change at Day 14 of Cycle 1 | 0.12 (1.064) | -0.01 (1.031)
  Change at Day 14 of Cycle 2 | 0.37 (1.293) | 0.03 (0.980)
  Change at Overall Day 56 | 0.43 (1.278) | 0.23 (1.528)

15. Secondary Outcome: Change From Baseline in the CF-Related Symptom Scores, as Assessed Using a Participant-Reported Questionnaire at Day 14 of Cycles 1 and 2 and Overall Day 56
Description: The CF symptom questionnaire includes questions related to daytime cough, nighttime cough, sputum volume, sputum clearance, physical fatigue, and shortness of breath. The participants (or their guardians) completed the CF symptom questionnaire, under the Investigator's supervision, before the TEPD, nasal mucosal curettage, pulmonary function tests, or sputum induction procedures were performed. For each symptom, the participants were asked to choose the response that best matched their experience during the 3 days before the questionnaire was completed. The scale of the 4 possible responses for each question was 0 (best response) to 4 (worse response). The sum of the scores for all of the questions was calculated. The scale for the sum of the scores was 0 (best response) to 24 (worse response). Overall Baseline data for the study and change from overall Baseline data at Day 14 of Cycles 1 and 2 and at overall Day 56 are presented.
Time Frame: Overall Baseline, Day 14 of Cycle 1 and Cycle 2 (1 cycle=28 days), and Overall Day 56
Population: All randomized participants who received at least 1 dose of study drug and had evaluable CF-related symptom scores.
Measure: Median (Full Range); unit: scores on a scale
Arm/Group | Ataluren 4, 4, and 8 mg/kg, Then Ataluren 10, 10, and 20 mg/kg | Ataluren 10, 10, and 20 mg/kg, Then Ataluren 4, 4, and 8 mg/kg
Number analyzed (Participants) | 15 | 15
scores on a scale
  Overall Baseline | 14.0 [7 to 19] | 11.0 [7 to 17]
  Change at Day 14 of Cycle 1: number analyzed (Participants) | 14 | 15
  Change at Day 14 of Cycle 1 | -0.5 [-7 to 6] | 0 [-5 to 4]
  Change at Day 14 of Cycle 2: number analyzed (Participants) | 15 | 14
  Change at Day 14 of Cycle 2 | -1.0 [-5 to 7] | 1.0 [-5 to 8]
  Change at Overall Day 56 | -1.0 [-7 to 9] | 0 [-6 to 8]

16. Secondary Outcome: PK: Area Under the Concentration Time Curve From Time 0 (Dosing) to 24 Hours (AUC0-24) of Ataluren
Description: All PK parameters were calculated using the actual postdose blood sampling times in relationship to the time of the first dose (morning dose) on Day 14 of each treatment cycle. AUC0-24 values were calculated by WinNonlin by extrapolation to 24 hours if the last sampling timepoint was before 24 hours and by interpolation if the last sampling timepoint was after 24 hours. Extrapolation of AUC to 24 hours was performed only if the last sampling timepoint did not deviate from the nominal collection time by more than approximately 10%.
Time Frame: 0 (predose), 2 and 3 hours postdose of the morning dose; 0 (predose), 2 and 3 hours postdose of the midday dose; and 0 hours (predose), 2, 3, and 12 hours postdose of the evening dose on Day 14 of Cycle 1 and Cycle 2
Population: All randomized participants who received at least 1 dose of study drug and had evaluable AUC0-24 data. The data for each dose level represents pooled data for participants in the low-to-high dose sequence and the high-to-low dose sequence.
Measure: Mean (Standard Error); unit: microgram*hours/milliliter (μg*h/mL)
Arm/Group | Ataluren 4, 4, and 8 mg/kg, Then Ataluren 10, 10, and 20 mg/kg | Ataluren 10, 10, and 20 mg/kg, Then Ataluren 4, 4, and 8 mg/kg
Number analyzed (Participants) | 30 | 30
microgram*hours/milliliter (μg*h/mL) | 121.52 (9.79) | 348.75 (21.46)

17. Secondary Outcome: Compliance With Study Treatment
Description: For each participant, compliance was described in terms of the percentage of drug actually taken relative to the amount that was prescribed (taking into account physician-prescribed reductions and interruptions). The number of doses described as "taken less than planned" includes cases in which the participants took less than the prescribed dose and/or cases in which the Investigator reduced the dose.
Time Frame: Baseline up to Day 14 in Cycle 1 and Cycle 2
Population: All randomized participants who received at least 1 dose of study drug and had evaluable compliance data. The data for each dose level represents pooled data for participants in the low-to-high dose sequence and the high-to-low dose sequence.
Measure: Median (Full Range); unit: percentage of doses
Arm/Group | Ataluren 4, 4, and 8 mg/kg, Then Ataluren 10, 10, and 20 mg/kg | Ataluren 10, 10, and 20 mg/kg, Then Ataluren 4, 4, and 8 mg/kg
Number analyzed (Participants) | 30 | 30
percentage of doses
  Percentage of doses taken as planned | 97.50 [81.8 to 100.0] | 100.0 [65.1 to 100.0]
  Percentage of doses missed | 2.40 [0 to 15.8] | 0 [0 to 16.2]
  Percentage of doses taken less than planned | 0 [0 to 10.5] | 0 [0 to 30.2]
  Percentage of doses taken greater than planned | 0 [0 to 0] | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: Overall Baseline up to Overall Day 56
Description: The data for each dose level represents pooled data for participants in the low-to-high dose sequence and the high-to-low dose sequence.
Groups:
- Ataluren 4, 4, and 8 mg/kg: Participants received ataluren at 4 milligrams in the morning, 4 mg/kg at midday, and 8 mg/kg in the evening for 14 days, followed by a 14-day follow-up period without treatment.
- Ataluren 10, 10, and 20 mg/kg: Participants received ataluren at 10 mg/kg in the morning, 10 mg/kg at midday, and 20 mg/kg in the evening for 14 days, followed by a 14-day follow-up period without treatment.
Arm/Group | Ataluren 4, 4, and 8 mg/kg | Ataluren 10, 10, and 20 mg/kg
Serious Adverse Events (participants affected / at risk) | 1/30 | 1/30
Other Adverse Events (participants affected / at risk) | 19/30 | 24/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ataluren 4, 4, and 8 mg/kg (N=30) | Ataluren 10, 10, and 20 mg/kg (N=30)
Cystic fibrosis pulmonary exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ataluren 4, 4, and 8 mg/kg (N=30) | Ataluren 10, 10, and 20 mg/kg (N=30)
Abdominal pain (Gastrointestinal disorders) | 6 | 8
Diarrhoea (Gastrointestinal disorders) | 3 | 2
Nausea (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Chest pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 2
Nasopharyngitis (Infections and infestations) | 1 | 1
Rhinitis (Infections and infestations) | 7 | 7
Stenotrophomonas infection (Infections and infestations) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Cystic fibrosis pulmonary exacerbation (Respiratory, thoracic and mediastinal disorders) | 4 | 6
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 0 | 2
Fatigue (General disorders) | 0 | 1
Thirst (General disorders) | 0 | 1
Laryngitis (Infections and infestations) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the Principal Investigator is that the Sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is up to 180 days from the time submitted to the sponsor for review. The sponsor may consult with the PI to require changes to the communication embargo.